CLINICAL TRIAL: NCT03380663
Title: Conditioning Based Intervention Strategies - ConBIS. A Research Study on the Potential of Remote Conditioning for Activation of Endogenous Organ Protection and the Underlying Molecular Mechanisms
Brief Title: Conditioning Based Intervention Strategies
Acronym: ConBIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ConBIS
Record Dates: First submitted 2017-08-23; First posted 2017-12-21 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-08

CONDITIONS: Ischemic Preconditioning
Keywords: blood flow restricted resistance exercise; remote ischemic conditioning; miRNA

STUDY DESIGN:
Intervention Model Description: A multi-center randomized control study, including single-treatment and repeated treatment trials on individuals suffering from heart failure and healthy control subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- RIC - Healthy (Active Comparator): Healthy subjects undergoing Remote Ischemic Conditioning (RIC) by inducing 3 or 4 five-minute cycles of limb ischemia and reperfusion using a tourniquet.
  Interventions: Procedure: Remote Ischemic Conditioning (RIC)
- RIC - HF (Active Comparator): Heart failure patients undergoing Remote Ischemic Conditioning (RIC) by inducing 3 or 4 five-minute cycles of limb ischemia and reperfusion using a tourniquet.
  Interventions: Procedure: Remote Ischemic Conditioning (RIC)
- BFRE - Healthy (Active Comparator): Healthy subjects undergoing low intensity blood flow restricted resistance exercise (BFRE) conducting 4 sets of bilateral knee extensions at 30% of 1RM until concentric contraction failure. The sets are intercepted by 30 seconds of rest (during rest the cuff's are still inflated).
  Interventions: Procedure: Remote Ischemic Conditioning (RIC)
- BFRE - HF (Active Comparator): Heart failure patients undergoing low intensity blood flow restricted resistance exercise (BFRE) conducting 4 sets of bilateral knee extensions at 30% of 1RM until concentric contraction failure. The sets are intercepted by 30 seconds of rest (during rest the cuff's are still inflated).
  Interventions: Procedure: Remote Ischemic Conditioning (RIC)
- TRT - Healthy (Active Comparator): Healthy subjects undergoing heavy intensive resistance training (TRT) undergoing 4 sets of 10-12 repetitions are performed in the knee extensor machine - load equaling 15RM and rest for 3 minutes).
  Interventions: Procedure: Remote Ischemic Conditioning (RIC)
- Control - Healthy (No Intervention): No intervention.
- Control - HF (No Intervention): No intervention.

INTERVENTIONS:
Procedure: Remote Ischemic Conditioning (RIC) — Remote Ischemic Conditioning (RIC) is a new treatment modality to attenuate reperfusion injury. Organ protection by RIC can be achieved simply by inducing 3 or 4 five-minute cycles of limb ischemia and reperfusion using a tourniquet or simple blood pressure cuff Ischemic resistance exercise training conducted as low-intensity blood flow restricted resistance exercise (BFRE), with a low occlusion pressure stimulus, which only compromises venous but not arterial blood flow. Much like RIC, BFRE is conducted as 3-5 cycles (sets of exercise) interspaced by short duration of recovery.
  High intensity traditional resistance training (TRT) is performed by sets of 10-12 repetitions are performed in the knee extensor machine - load equaling 15RM and rest for 3 minutes).
  Other Names: Blood Flow Restricted resistance Exercise (BFRE); Traditional Resistance Training (TRT)
  Arms: BFRE - HF; BFRE - Healthy; RIC - HF; RIC - Healthy; TRT - Healthy

SUMMARY:
The overall objective of this study is to uncover and utilize the mechanisms behind the activation of endogenous organ protection by remote ischemic conditioning (RIC), high intensity traditional resistance training (TRT) and low intensity blood flow restricted resistance exercise (BFRE) with the perspective of defining their applicability for immediate organ protection in ischemia-reperfusion injury (acute conditioning) and subsequent tissue repair (chronic conditioning) during a prolonged recovery period. This objective will be achieved by studying which and how molecular pathways underlying these protective mechanisms are shared and can be transferred to treat medical conditions. A specific focus is the roles of EVs and miRNAs. Another objective is to explore how exercise training with and without ischemia can counteract muscle wasting.

DETAILED DESCRIPTION:
Background

Clinical background - ischemia related and inflammatory conditions The pandemic of cardiovascular disease has immense negative effects on global population health and life expectancy. The most detrimental acute ischemic events are myocardial infarction and stroke. Organ failure caused by ischemia-reperfusion syndromes such as stroke and myocardial infarction constitutes the leading cause of death globally and carry a vast socio-economical burden. Overall, 17 million people worldwide are estimated to die from cardiovascular diseases (7.4 million from ischemic heart disease and 6.7 million from stroke). Attempts to modify risk factor and life style related growth in cardiovascular disease are important and have been successful in some parts of the world, but improved treatment of acute and chronic cardiovascular disease is crucial to alleviate the disease burden.

In acute ischemic conditions such as myocardial infarction and stroke, early and successful restoration of tissue perfusion following an ischemic event is the most effective strategy to reduce tissue injury and improve clinical outcome, but reperfusion may induce further tissue damage itself, so-called reperfusion injury. Although reperfusion strategies continue to progress with improved logistics and medical treatment, even optimal acute reperfusion treatment may leave patients with chronic ischemic disease. Actually, as initial survival has improved due to improvements in acute reperfusion therapy, the number of patients with chronic ischemic heart disease is growing globally (more than 35 million people worldwide suffering from heart failure). Collectively, patients with heart failure have a poorer 5-year survival rate than patients with most types of cancer. However, the development of effective drugs to target the detrimental effects of reperfusion injury itself has proven to be a challenge. Several pharmacologic strategies showing convincing effects in animal models of ischemia-reperfusion injury have failed to translate into clinical benefit.

A key feature of heart failure caused by chronic ischemic heart disease is inflammation, which shares mechanisms with other inflammatory conditions such as inflammatory bowel disease and ankylosing spondylitis. Further debilitating, heart failure also exerts a negative effect on habitual physical activity and skeletal muscle tissue health, producing multiple detrimental effects on whole-body metabolism and mobility. A common underlying mechanistic trait of these processes could be regulation by circulating small non-coding RNAs (micro RNAs or miRNAs/miRs).

Scientific background Remote ischemic conditioning The main prognostic determinant of outcome in acute myocardial infarction is the extent of tissue damage (infarct size), which is determined not only by the duration of ischemia but also by injury caused by reperfusion injury. Remote Ischemic Conditioning (RIC) is a new treatment modality to attenuate reperfusion injury. Organ protection by RIC can be achieved simply by inducing 3 or 4 five-minute cycles of limb ischemia and reperfusion using a tourniquet or simple blood pressure cuff. With few exceptions, RIC has consistently been shown to exert powerful protection against ischemia-reperfusion injury in the heart, brain, kidneys, lungs, and liver in animal models, and RIC has successfully been translated into clinical use. A specific advantage of RIC is its easy applicability during ongoing ischemia of the target organ, which has been exploited in animal models and humans to show that RIC reduces injury during evolving myocardial infarction and stroke.

While the mediators and mechanisms of RIC remain to be identified, RIC has been shown to 1) induce cytoprotection, 2) improve endothelial function and microcirculation, and 3) modify inflammation - all three key players in the pathology behind heart failure - suggesting a potentially powerful tool to simultaneously counteract detrimental biological processes involved in the development of heart failure. RIC may have further potential because continued RIC after myocardial infarction seems to induce sustained benefits during the following adverse remodeling of the heart. The anti-inflammatory effects may be of importance in other conditions involving acute or chronic inflammation.

Ischemia and conditioning with blood flow restricted resistance exercise Exercise is traditionally categorized and practiced as either oxygen-demanding aerobic endurance exercise with effect on metabolic properties or mechanically stressing resistance exercise with effect on contractile properties. In addition to local myocellular effects, exercise appears to promote molecular inter-organ communication. Indeed, recent studies have demonstrated the ability of traditional exercise regimens to protect against e.g. myocardial ischemia-reperfusion injury and also to improve cognitive function, hence the conception that "exercise is medicine". Studies suggest that these remote effects are induced by myocellular production of circulatory mediators to influence tissues of remote organs. Exercise-induced muscle-organ cross-talk may, similar to RIC, rely on extracellular vesicle derived miRNA (see next paragraph). Supporting such a notion, is the finding that high intensity traditional resistance exercise evokes increased transcription of miR133b, since miR133b has recently been demonstrated to promote recovery after stroke via transfer of exosome-enriched extracellular particles. However, high intensity traditional exercise can produce muscle injury and may therefore not comply with exercise in patients with cardiovascular or other chronic muscle wasting diseases.

A novel approach may be offered by Ischemic resistance exercise training conducted as low-intensity blood flow restricted resistance exercise (BFRE), with a low occlusion pressure stimulus, which only compromises venous but not arterial blood flow. Much like RIC, BFRE is conducted as 3-5 cycles (sets of exercise) interspaced by short duration of recovery. By this mechanically very gentle approach, muscle accretion similar to that of high intensity traditional resistance training (TRT) can be achieved, possibly due to acceleration of metabolic build-up or activation of muscle stem cells. Interestingly, new results by us, demonstrate that BFRE can mediate long-lasting preconditioning effects in muscle. Since low-intensity BFRE mimics events of both traditional high intensity resistance exercise (occlusion-reperfusion) and traditional aerobe exercise (hypoxia), BFRE can be speculated to drive health beneficial metabolic as well as anabolic adaptations in the muscle. Based on its resemblance to RIC, BFRE likely also affect remote tissues and infer remote organ protection. The extent to which RIC and exercise regimens may share or overlap or differ mechanistically - and potentially exert additive effects - is unknown, but application of BFRE entails highly promising clinical perspectives.

Micro RNA signaling Circulating extracellular vesicles (EVs) are small particles released from plasma membranes from almost all cell types. These EVs seem to act as transport systems in the body carrying a cargo of signaling substances including miRNAs. miRNAs are also effector molecules in ischemic events, e.g. myocardial miRNA144 (miR144) levels are reduced by ischemic reperfusion injury (IR injury), which is attenuated by RIC. RIC also induces increased circulatory EV levels, while EVs enriched with miR22 and miR451 from anoxic cultured MSCs and cardiomycyte progenitor cells mitigate cardiac injury. Potentially, treatment with specific miRNA loaded into EVs may provide protection against acute and chronic effects of myocardial ischemia-reperfusion injury in patients [19]. EVs are also believed to contain other substances including anti-inflammatory components acting in synergy with miRNA to exert the full effect of the signaling cascade.

Objectives The overall objective of this study is to uncover and utilize the mechanisms behind the activation of endogenous organ protection by remote ischemic conditioning (RIC), high intensity traditional resistance training (TRT) and low intensity blood flow restricted resistance exercise (BFRE) with the perspective of defining their applicability for immediate organ protection in ischemia-reperfusion injury (acute conditioning) and subsequent tissue repair (chronic conditioning) during a prolonged recovery period. This objective will be achieved by studying which and how molecular pathways underlying these protective mechanisms are shared and can be transferred to treat medical conditions. A specific focus is the roles of EVs and miRNAs. Another objective is to explore how exercise training with and without ischemia can counteract muscle wasting.

Hypotesis

The overall hypothesis of the proposal is that RIC and exercise potentiated by BFRE and TRT release circulating protective mediators that exert immediate protective effects against IR injury as well as promote beneficial repair during subsequent tissue rebuilding and in chronic inflammatory conditions. Specifically, we will test the following hypotheses:

1. RIC, BFRE and TRT share organ protecting and anti-inflammatory properties induced through common miRNA signaling pathways
2. Long lasting effect of RIC, BFRE and TRT can be achieved by repeated treatment, and the chronic effects include anti-inflammatory and anti-ischemic properties of clinical relevance by:

   1. Improving ventricular function and reduce symptoms in patients with heart failure and chronic ischemic heart disease (individual sub-study, a separate application has been submitted to and approved by De Videnskabsetiske Komitéer).
   2. Counteracting muscle wasting in patients with heart failure.
3. BFRE is a more effective mean to increase muscle mass, muscle power and muscle function compared to TRT.
4. Non-conditioned EVs can be loaded with RIC, BFRE and specific miRNA, in vitro and exert immediate protective effects against IR injury upon intravenous injection (future sub-study)

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the written and spoken information and to give informed consent for inclusion.
* Age between 18 and 80 years
* Able to sit in a knee extension machine
* Able to deliver muscle biopsies
* Able to train 3 times per week during a 6-week period

Inclusion Criteria - heart failure patients

* Chronic congestive ischemic heart failure
* LV ejection fraction ≤45%
* NYHA function class II-IV

Inclusion Criteria - healthy subjects

• See general criteria for inclusion

Exclusion Criteria - healthy subjects

* Myocardial infarction
* Angina pectoris

Exclusion Criteria:

* Pregnancy
* Diabetes mellitus
* Peripheral neuropathy
* Dialysis treatment
* Severe peripheral arterial disease
* Concomitant acute life threatening medical condition
* Medications known to modify the effect of ischemic conditioning such as cyclosporin and glibenclamide.
* Recent cardiovascular hospitalization (within last 30 days)
* Intracranial aneurisms, arteriovenous malformation, cerebral neoplasm or abscess.
* Myocardial infarction
* Angina pectoris
* Severe arterial hypertension (≥ 180/≥ 110 mmHg) or moderate arterial hypertension (160-179/100-109) despite medical treatment.
* Moderate to severe cardiac valve disease
* Beta blocker medication
* Moderate or severe chronic obstructive pulmonary disease
* Decreased kidney function - eGFR < 60 ml/min.

Criteria for stopping the intervention or investigations

* Severe discomfort and/or by request of the participant.
* Safety considerations as assessed by the investigator.
* Withdrawal of informed consent.
* Not able to fulfill the protocol.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Changes in miRNA and EV content in blood samples | 6 Weeks
  Analyzing miRNA sequences

SECONDARY OUTCOMES:
Effects on muscle endurance | 6 weeks
  Number of repetitions in curl machine and mitochondrial oxidative capacity
Effects on inflammatory state | 6 weeks
  Changes in cytokines
Changes in skeletal muscle myofibrillar and mitochondrial protein synthesis | 6 weeks
  Histochemical examination
Protection against IR injury in isolated rat/rabbit hearts and isolated cells | 6 weeks
  Histological examination
Changes in skeletal muscle growth and strength | 6 weeks
  Muscle strength measurement - force

CONTACTS AND LOCATIONS:
Overall Officials: Hans Erik Bøtker, MD, PhD, Study Director — Department of Clinical Medicine, Department of Cardiological Medicine, Aarhus University Hospital
Locations (1):
- Aarhus University, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lassen TR, Just J, Hjortbak MV, Jespersen NR, Stenz KT, Gu T, Yan Y, Su J, Hansen J, Baek R, Jorgensen MM, Nyengaard JR, Kristiansen SB, Drasbek KR, Kjems J, Botker HE. Cardioprotection by remote ischemic conditioning is transferable by plasma and mediated by extracellular vesicles. Basic Res Cardiol. 2021 Mar 10;116(1):16. doi: 10.1007/s00395-021-00856-w. PMID 33689033
- [Derived] Groennebaek T, Sieljacks P, Nielsen R, Pryds K, Jespersen NR, Wang J, Carlsen CR, Schmidt MR, de Paoli FV, Miller BF, Vissing K, Botker HE. Effect of Blood Flow Restricted Resistance Exercise and Remote Ischemic Conditioning on Functional Capacity and Myocellular Adaptations in Patients With Heart Failure. Circ Heart Fail. 2019 Dec;12(12):e006427. doi: 10.1161/CIRCHEARTFAILURE.119.006427. Epub 2019 Dec 13. PMID 31830830